CLINICAL TRIAL: NCT02473094
Title: Metformin in Association to Chemoradiotherapy for the Neoadjuvant Treatment of Locally Advanced Rectal Cancer: a Randomized, Placebo-controlled Phase II Study
Brief Title: Neoadjuvant Metformin in Association to Chemoradiotherapy for Locally Advanced Rectal Cancer
Acronym: NEOMETRE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Ligia Traldi Macedo, Clinical Oncology, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEOMETRE201501
Record Dates: First submitted 2015-06-13; First posted 2015-06-16 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Rectal Neoplasms; Adenocarcinoma; Carcinoma
Keywords: Metformin; Rectal Cancer; Rectum; Radiotherapy; Capecitabine; Neoadjuvant; Adenocarcinoma; Carcinoma
MeSH Terms: conditions — Rectal Neoplasms; Adenocarcinoma; Carcinoma | interventions — Capecitabine; Metformin; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neoadjuvant capecitabine and metformin (Experimental): * Capecitabine 825 mg/m2 bid D1-5, q7d, for five weeks;
  * Metformin 2500mg/d for five weeks;
  * 3D radiotherapy 50,4Gy divided in 25 fractions
  Interventions: Drug: Capecitabine; Drug: Metformin; Radiation: Radiotherapy
- Neoadjuvant capecitabine and placebo (Placebo Comparator): * Capecitabine 825 mg/m2 bid D1-5, q7d, for five weeks;
  * Placebo 2500mg/d for five weeks;
  * 3D radiotherapy 50,4Gy divided in 25 fractions
  Interventions: Drug: Capecitabine; Radiation: Radiotherapy; Drug: Placebo

INTERVENTIONS:
Drug: Capecitabine — Capecitabine 825mg/m2 bid, D1-D5 q7d
  Other Names: Xeloda
Drug: Metformin — Metformin up to 2500mg/d
  Other Names: Glifage, Dimefor, Glucoformin, Glucophage
  Arms: Neoadjuvant capecitabine and metformin
Radiation: Radiotherapy — 3D radiotherapy 50,4Gy divided in 25 fractions
  Other Names: RDT
Drug: Placebo — Placebo up to 2500mg/d
  Arms: Neoadjuvant capecitabine and placebo

SUMMARY:
A phase II, randomized study of placebo versus metformin in association to chemotherapy with capecitabine and radiation in the neoadjuvant treatment of locally advanced (T3-4N0M0 or TxN1-2M0) rectal carcinomas.

DETAILED DESCRIPTION:
NEOMETRE is a randomized, double blind trial aiming to evaluate the efficacy and tolerability of metformin in association to chemoradiotherapy for the preoperative treatment of locally advanced (T3-4N0M0 or TxN1-2M0) rectal carcinomas.

Patients eligible for this study will be submitted to neoadjuvant 3D radiotherapy with 50,4 Gray (Gy) divided in 25 applications, in association to capecitabine, 825mg/m2 bid for five days every week. The participants will be randomized to daily metformin or placebo during the chemoradiotherapy period. The primary end-point is pathological complete response. The secondary end-points are recurrence-free survival (RFS), disease-free survival (DFS), overall survival (OS), local recurrence rate, overall response rate, sphincter preservation rate, quality of life (QoL) and toxicity.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older;
* biopsy proven poorly differentiated carcinoma or adenocarcinoma of the rectum;
* lesions located within 12 cm of the anal verge (from colonoscopy assessment);
* ability to tolerate oral treatment;
* locally advanced tumor, classified by the presence of positive regional lymph nodes or primary tumor invasion beyond the serosa (T3 or T4), assessed by MRI;
* eligibility for curative surgery (no distant metastasis or invasion of bony structures of the pelvis);
* Performance Status (PS) Eastern Cooperative Oncology Group (ECOG) 0-2;
* adequate hematologic functions (hemoglobin ≥ 10 g / dL [5.6 mmol / L]; neutrophil count ≥ 1,500 / mm3 and platelet count ≥ 100,000 / mm3), adequate renal function (serum creatinine less than 1.5 times the UNL) and adequate hepatic function (bilirubin less than 1.5 times the UNL; aspartate aminotransferase and alanine aminotransferase less than 2.5 times the UNL);

Exclusion Criteria:

* known hypersensitivity to metformin or its excipients;
* squamous carcinomas of the rectum or anal canal;
* chronic treatment with corticosteroids or other immunosuppressive agents;
* treatment with oral antidiabetic products;
* distant metastasis at diagnosis or tumor invasion of pelvic bone structures that may proscribe curative intent surgery;
* chronic or acute infections;
* use of drugs under study up to four weeks prior to randomization;
* pregnant or nursing patients;
* prior radiotherapy to the pelvic region;
* myocardial infarction up to six months prior to randomization, or uncontrolled ischemic heart disease;
* congestive heart insufficiency New York Heart Association (NYHA) III-IV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Pathological Complete Response | 8 to 16 weeks after neoadjuvant treatment completion
  Pathological evaluation of the surgical specimen. Complete response will be defined as absence of neoplastic tissue upon pathological exam.

SECONDARY OUTCOMES:
Overall Response Rate | 4 to 6 weeks after neoadjuvant treatment completion
  Magnetic Resonance Imaging (MRI) assessment to compare the response of chemoradiotherapy+metformin versus chemoradiotherapy+placebo.
Sphincter Preservation Rate | 8 to 16 weeks after neoadjuvant treatment completion
  Rate of anal sphincter preservation during curative intent surgery.
Toxicity will be assessed using National Cancer Institute Common Toxicity Criteria for Adverse Effects (NCI CTCAE) v4.03 | up to 4 weeks after neoadjuvant treatment completion
  Safety and tolerability will be assessed using National Cancer Institute Common Toxicity Criteria for Adverse Effects (NCI CTCAE) v4.03. The number of patients in each arm experiencing grade 3-5 adverse events ou AE (for each AE) over the total number of subjects will be measured, and the proportion of patients experiencing AE in each arm will be compared using uncorrected chi-square test. AE will be recorded in baseline and in each visit, and the worst grade AE will be considered.
Local Recurrence Rate | up to 5 years
  Rate of local or pelvic recurrence during follow up.
Local Recurrence Free Survival | up to 5 years
  The number of subjects without local relapse will be measured 6mo after the start of therapy, also after 1, 3 and 5 years from the start of therapy. Local recurrence free survival will be analysed with log-rank test, and reported as Hazard Ratio (HR) with respective 95% Confidence Interval (CI) and p value, and its median value will be estimated with kaplan-meyer method.
Disease Free Survival | up to 5 years
  The number of subjects without relapse will be measured 6mo after the start of therapy, also after 1, 3 and 5 years from the start of therapy. Disease free survival will be analysed with log-rank test, and reported as HR with respective 95% CI and p value, and its median value will be estimated with kaplan-meyer method.
Overall Survival | up to 5 years
  The number of subjects without death (any cause) will be measured 6mo after the start of therapy, and also after 1, 3 and 5 years from the start of therapy. Overall survival will also be analysed with log-rank test, and reported as HR with respective 95% CI and p value, and median OS will be estimated with kaplan-meyer method. All calculations will be performed 6 months after the last patient recruited. Also, the survival rate at year one, three and five will be calculated.
Quality of Life | up to 20 weeks after neoadjuvant treatment completion
  European Organization for Research and Treatment of Cancer Quality of Life Questionaire (EORTC QLQ)-C30 and EORTC QLQ-CR29 will be assessed on screening, at the last day of neoadjuvant treatment, 4 weeks after neoadjuvant treatment completion and up to 4 weeks after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ligia T Macedo, MD, Principal Investigator — Clinical Oncology Department, State University of Campinas (UNICAMP); Jose BC Carvalheira, MD, PhD, Study Chair — Clinical Oncology Department, State University of Campinas (UNICAMP)
Locations (1):
- Clinical Oncology Department - General Hospital - State University of Campinas (UNICAMP), Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No